CLINICAL TRIAL: NCT04599556
Title: Clinical Trial for the Safety and Efficacy of Anti-CD7 Chimeric Antigen Receptor Cell Therapy for Patients With Relapsed or Refractory CD7 Positive Hematological Malignancy
Brief Title: Clinical Trial for the Safety and Efficacy of Anti-CD7 CAR-T Cell Therapy for Patients With Relapsed or Refractory CD7 Positive Hematological Malignancy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD7-001
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: CD7+ Acute Leukemia; CD7+ Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T-ALL/LBL (Experimental)
  Interventions: Biological: anti-CD7 CAR-T
- T-NHL (Experimental)
  Interventions: Biological: anti-CD7 CAR-T
- AML (Experimental)
  Interventions: Biological: anti-CD7 CAR-T

INTERVENTIONS:
Biological: anti-CD7 CAR-T — Lymphodepleting chemotherapy followed by anti-CD7 CAR-T infusion

SUMMARY:
This is a prospective, open-label, single-center clinical trial. This study will evaluate the safety and efficacy of anti-CD7 CAR-T cells in the treatment of relapsed or refractory CD7 positive T-ALL/LBL, T-NHL and AML. The primary endpoints are dose limiting toxicity (DLT) and the incidence of treatment emergent adverse event (TEAE).

ELIGIBILITY:
Inclusion Criteria:

1. Total bilirubin ≤ 51 μmol / L, ALT and AST ≤ 3 times of the upper limit of normal value, serum creatinine ≤ 176.8 μmol / L;
2. Echocardiography shows left ventricular ejection fraction (LVEF) ≥ 50%;
3. There is no active pulmonary infection, and the oxygen saturation during air inhalation is more than 92%;
4. The estimated survival time is more than 3 months;
5. ECOG score was 0-2;
6. The patients or their legal guardians voluntarily participated in the trial and signed the informed consent.

For T-ALL/LBL:

1. Patients is histologically diagnosed with CD7 Positive T-ALL/LBL according to the Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (ALL) (2020. V1) by National Comprehensive Cancer Network (NCCN).
2. The diagnosis is consistent with r/r CD7 + T-ALL/LBL, and includes any of the following conditions:

   1. No CR was obtained by standard chemotherapy;
   2. The first induction was CR, but the duration of CR was less than 12 months;
   3. No CR was obtained after the first or multiple remedial treatment;
   4. Relapse twice or more;
3. The number of blast cells in bone marrow was more than 5% (morphology) and / or > 1% (flow cytometry).

For T-NHL:

1. Patients is histologically diagnosed with CD7 Positive T-NHL according to The 2016 revision of the World Health Organization classification of lymphoid neoplasms.
2. r/r T-NHL, and includes any of the following conditions:

   1. No response or relapse after second or more lines of chemotherapy;
   2. Primary refractory ot chemotherapy;
   3. Relapse after autologous stem cell transplantation;
3. According to the Lugano 2014 criteria, there is at least one evaluable tumor lesion.

For AML:

1. Patients is histologically diagnosed with CD7 Positive AML according to the Clinical Practice Guidelines for Acute Myeloid Leukemia (AML) (2020. V3) by National Comprehensive Cancer Network (NCCN).
2. The diagnosis is consistent with r/r CD7 + AML, and includes any of the following conditions:

   1. No CR was obtained by standard chemotherapy;
   2. The first induction was CR, but the duration of CR was less than 12 months;
   3. No CR was obtained after the first or multiple remedial treatment;
   4. Relapse twice or more;
3. The number of blast cells in bone marrow was more than 5% (morphology) and / or > 1% (flow cytometry).

Exclusion Criteria:

1. Patients with history of epilepsy or other central nervous system diseases;
2. Patients with prolonged QT or severe heart disease;
3. Pregnant or lactating women (the safety of this therapy for unborn children is unknown);
4. The patients with uncontrolled active infection;
5. Active hepatitis B or hepatitis C virus infection;
6. Previous application of gene therapy;
7. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
8. Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0mg/dl;
9. Those who suffer from other uncontrolled diseases are not suitable to join the study;
10. HIV infection;
11. Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | 28 days
Treatment Emergent Adverse Event | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Y, Zhang M, Yang T, Mo Z, Wei G, Jing R, Zhao H, Chen R, Zu C, Gu T, Xiao P, Hong R, Feng J, Fu S, Kong D, Xu H, Cui J, Huang S, Liang B, Yuan X, Cui Q, Guo H, Yu Y, Feng Y, Jin C, Ren J, Chang AH, Wang D, Huang H. Sequential CD7 CAR T-Cell Therapy and Allogeneic HSCT without GVHD Prophylaxis. N Engl J Med. 2024 Apr 25;390(16):1467-1480. doi: 10.1056/NEJMoa2313812. PMID 38657244
- [Derived] Xu X, Zu C, Zhang M, Xiao P, Hong R, Feng J, Xu H, Cui J, Yu J, Shi J, Wei G, Chang AH, Huang H, Hu Y. HLA Fully-Mismatched Sibling-Derived CD7 CAR-T Therapy Bridging to Haploidentical Hematopoietic Stem Cell Transplantation for Hepatosplenic gammadelta T-cell Lymphoma. Cell Transplant. 2023 Jan-Dec;32:9636897231194265. doi: 10.1177/09636897231194265. PMID 37667507